CLINICAL TRIAL: NCT05666128
Title: A Multi-center, Double-blind, Randomized, Placebo-controlled, Parallel-group, Phase 2 Study to Assess the Efficacy and Safety of HD-6277 in Adult Patients with Inadequate Control of Type 2 Diabetes Mellitus by Diet and Exercise
Brief Title: Efficacy and Safety of HD-6277 in Adult Patients with Inadequate Control of Type 2 Diabetes Mellitus by Diet and Exercise
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hyundai Pharm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HT-006-02
Record Dates: First submitted 2022-12-18; First posted 2022-12-27 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- HD-6277 100mg (Experimental)
  Interventions: Drug: HD-6277
- HD-6277 50mg (Experimental)
  Interventions: Drug: HD-6277
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HD-6277 — HD-6277 100mg
  Arms: HD-6277 100mg
Drug: HD-6277 — HD-6277 50mg
  Arms: HD-6277 50mg
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
A Multi-center, Double-blind, Randomized, Placebo-controlled, Parallel-group, Phase 2 Study to Assess the Efficacy and Safety of HD-6277 in Adult Patients With Inadequate Control of Type 2 Diabetes Mellitus by Diet and Exercise

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of T2DM with HbA1c between 7.0% and 10.0% (inclusive) while on diet and exercise alone for at least 6 weeks prior to screening.

Exclusion Criteria:

* Type 1 diabetes or another immune-mediated diabetes syndrome

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2022-06-17 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2023-07-28 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c(%) at weeks 12 from baseline | at weeks 12 from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Included Severance Hospital, 10 sites, Seoul, South Korea